CLINICAL TRIAL: NCT04571151
Title: Efficacy and Safety of Sorilux in Maintenance Treatment of Moderate Type Plaque Psoriasis After Combination Treatment of Lexette and Sorilux for 2 Weeks
Brief Title: Efficacy and Safety of Sorilux in Maintenance Treatment of Moderate Type Plaque Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Skin Sciences, PLLC (Other)
Responsible Party: Principal Investigator, Leon H. Kircik, MD, Medical Director, Skin Sciences, PLLC
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LEX-2001
Record Dates: First submitted 2020-09-23; First posted 2020-09-30 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to study treatment at a 1:1 ratio: of Lexette plus Sorilux for 2 weeks versus Lexette plus vehicle for 2 weeks. Those subjects who are clear or almost clear at the end of 2 weeks will be re-randomized into Sorilux for 6 weeks versus vehicle for 6 weeks at 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. Medication's label will be covered. Only the study coordinator would be able to identify the medication.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lexette + Sorilux (Active Comparator): Halobetasol Propionate Topical Foam (Lexette Foam) + Calcipotriol Foam (Sorilux Foam) for 2 weeks
  Halobetasol Propionate Topical Foam (Lexette Foam) would be applied over the affected area twice daily for 2 weeks. Each gram of Halobetasol Propionate Topical Foam contains 0.5 mg of halobetasol propionate.
  Calcipotriol Foam (Sorilux Foam) would be applied over the affected area twice daily for 2 weeks 5 minutes after the Lexette application. SORILUX Foam contains calcipotriene 50 mcg/g.
  Interventions: Drug: LEXETTE 0.05% Topical Foam; Drug: Sorilux 0.005 % Topical Foam
- Lexette + Vehicle (Placebo Comparator): Halobetasol Propionate Topical Foam (Lexette Foam) + Vehicle Foam for 2 weeks
  Halobetasol Propionate Topical Foam (Lexette Foam) would be applied over the affected area twice daily for 2 weeks. Each gram of Halobetasol Propionate Topical Foam contains 0.5 mg of halobetasol propionate.
  Vehicle Foam would be applied over the affected area twice daily for 2 weeks 5 minutes after the Lexette application.
  Interventions: Drug: LEXETTE 0.05% Topical Foam; Other: Vehicle Foam
- Sorilux (Active Comparator): Calcipotriol Foam (Sorilux Foam) for 6 weeks
  Participants from Groups A and B who are clear or almost clear at the end of 2 weeks will be re-randomized into Groups 1 and 2.
  Calcipotriol Foam (Sorilux Foam) would be applied over the affected area twice daily for 6 weeks. SORILUX Foam contains calcipotriene 50 mcg/g.
  Interventions: Drug: Sorilux 0.005 % Topical Foam
- Vehicle (Placebo Comparator): Vehicle Foam for 6 weeks.
  Participants from Groups A and B who are clear or almost clear at the end of 2 weeks will be re-randomized into Groups 1 and 2.
  Vehicle Foam would be applied over the affected area twice daily for 6 weeks.
  Interventions: Other: Vehicle Foam

INTERVENTIONS:
Drug: LEXETTE 0.05% Topical Foam — Halobetasol Propionate Topical Foam (Lexette Foam) would be applied over the affected area twice daily for 2 weeks.
  Other Names: Halobetasol Propionate Topical Foam
  Arms: Lexette + Sorilux; Lexette + Vehicle
Drug: Sorilux 0.005 % Topical Foam — Calcipotriol Foam (Sorilux Foam) would be applied over the affected area twice daily for 2 weeks 5 minutes after the Lexette application. SORILUX Foam contains calcipotriene 50 mcg/g.
  Other Names: Calcipotriol Foam
  Arms: Lexette + Sorilux; Sorilux
Other: Vehicle Foam — Vehicle Foam would be applied over the affected area twice daily for 6 weeks.
  Arms: Lexette + Vehicle; Vehicle

SUMMARY:
The study seeks to show whether there is additional benefit of using Lexette and Sorilux in the beginning of the treatment, and then maintenance treatment of Sorilux alone in moderate plaque type psoriasis patients.

DETAILED DESCRIPTION:
This is a single-center, double-blind study. Approximately 30 qualified subjects will be enrolled into a 8 weeks study.

The study drugs that will be used in this study are Lexette® (0.05% Halobetasol propionate foam) and Sorilux® (calcipotriene foam). Both Lexette and Sorilux are approved by the United States Food and Drug Administration (FDA) to treat psoriasis.

Subjects will be randomized to study treatment at a 1:1 ratio: of Lexette plus Sorilux for 2 weeks versus Lexette plus vehicle for 2 weeks. Those subjects who are clear or almost clear at the end of 2 weeks will be re-randomized into Sorilux for 6 weeks versus vehicle for 6 weeks at 1:1 ratio.

Subjects will attend a Screening Visit/Baseline visit and if found eligible will be randomized to study treatment. Total study period is 8 weeks. Study visits will be, screening/baseline, week 2 and week 8. Study assessments will be at each visit: BSA, PGA, Itch VAS, DLQI, and TLSS in addition to standard medical assessments. There will be a standard prohibited medication/treatment and washout periods.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female subjects of any race, 18 years of age or higher. Female subjects of childbearing potential must have a (-)UPT result at within 7 days of the first dose of study drug and practice a reliable method of contraception throughout the study;

   A female is considered of childbearing potential unless she is:

   - postmenopausal > 5Y, without a uterus and/or both ovaries; or has been surgically sterile for > 6M.

   Reliable methods of contraception are:

   - hormonal methods or IUD in use > 90d prior to study drug administration, barrier methods plus spermicide in use > 14d prior, or vasectomized partner.

   [Exception: Female subjects of CBP who are not sexually active are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided they are counseled to remain sexually inactive for the duration of the study and understand the risks involved in getting pregnant during the study.]
2. Subjects with moderate plaque type psoriasis.
3. Physician Global Assessment (PGA) score of 3.
4. Able to understand study requirements and sign Informed Consent/HIPAA forms.
5. Target lesion must be at least 2cm in diameter

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control, or male subjects planning a pregnancy with their spouse or partner while in the study.
2. History of hypercalcemia or vitamin D toxicity or history of significant renal or hepatic disease
3. Patients with guttate, erythrodermic, or pustular psoriasis
4. Serious skin condition (other than psoriasis) or uncontrolled medical condition (in the opinion of the investigator).
5. Skin conditions (e.g. eczema) that may interfere with evaluations of psoriasis.
6. Known hypersensitivity to Lexette or Sorilux Foam or any of its components.
7. Current drug or alcohol abuse (Investigator opinion).
8. Subject unable to commit to all the assessments required by the protocol.
9. Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects who maintain clear or almost clear on Physician Global Assessment (PGA) at Week 8 | Week 8
  Physician assessment of disease severity. 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate

SECONDARY OUTCOMES:
Percent of subjects who maintain clear or almost clear on Physician Global Assessment (PGA) at Week 2 | Week 2
  Physician assessment of disease severity. 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate
Change in Visual Analogue Scale (VAS) at week 2 and week 8 | Screening/Baseline, Week 2, Week 8
  The VAS is a scale consisting of a 10cm long line and a single question used for measuring itch intensity. The left end point represents "no itch" and the right end point the "worst imaginable itch".
Change in Dermatology Life Quality Index (DLQI) at week 2 and week 8 | Screening/Baseline, Week 2, Week 8
  The Dermatology Life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question is scored on a four-point Likert scale:
  Very much = 3, A lot = 2, A little = 1, Not at all = 0, Not relevant = 0, Question unanswered = 0. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Change in Total Lesion Severity Score (TLSS) at week 2 and week 8 | Screening/Baseline, Week 2, Week 8
  A combined score of disease severity of target lesion which includes assessment of erythema (0=none, 2=pink, 4=red, 6=very red, 8=extremely red), induration (0=no evidence of plaque above normal skin level, 2=slight definite elevation above normal skin level, 4=moderate elevation with rounded or sloped edges to plaque, 6=marked elevation with hard sharp edges to plaque, 8=very marked elevation with very hard sharp edges to plaque), and scaling (0=no evidence of scaling on lesion, 2= mild mainly fine scales with some of lesion at least partially covered, 4=moderate somewhat coarser scale and most of lesion at least partially covered, 6= severe coarse thick scales and rough surface covering virtually all of lesion, 8=very severe coarse very thick scales and rough surface covering entire lesion)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H Kircik, Principal Investigator — Skin Sciences, PLLC
Locations (1):
- Skin Sciences, PLLC, Louisville, Kentucky, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT04571151/Prot_SAP_000.pdf